CLINICAL TRIAL: NCT05042024
Title: Supplementation With L-ornithine Increases Representation Density of CD68+ and CD163+ Macrophages in Human Periodontitis Gingiva and Can Modulate Macrophages Phenotypes. Randomized Controlled Pilot Trial
Brief Title: Supplementation With L-ornithine But Not L-arginine Increases Density of CD68+ and CD163+ Macrophages in Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ukrainian Medical Stomatological Academy (Other)
Responsible Party: Principal Investigator, Igor Kaydashev, Honored Master of Science and Technology of Ukraine, Doctor of Medical Sciences, Professor Vice-Rector for Research and Development, Ukrainian Medical Stomatological Academy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120U101151
Record Dates: First submitted 2021-08-31; First posted 2021-09-13 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Periodontitis
Keywords: L-arginine; L-ornithine; M1 M2 macrophages; macrophages-targeted therapy; periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Patients were grouped by stratified randomization into three groups: the SRP Group (patients received conventional periodontal therapy including scaling and root planing as a full-mouth procedure, n=25); the Arg Group (patients received oral L-arginine aspartate (Yuria-Pharm, Ukraine) at a dose of 1 g t.i.d. for 10 days after conventional periodontal therapy, n=25); and the Orn Group (patients received oral L-ornithine aspartate (Farmak, Ukraine) at a dose of 3 g t.i.d. for 15 days after conventional periodontal therapy, n=25).
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the SRP Group (Active Comparator): Patients received conventional periodontal therapy including scaling and root planing as a full-mouth procedure, n=25.
  Interventions: Procedure: Scaling and root planing
- the Arg Group (Experimental): Patients received oral L-arginine aspartate (Yuria-Pharm, Ukraine) at a dose of 1 g t.i.d. for 10 days after conventional periodontal therapy, n=25.
  Interventions: Procedure: Scaling and root planing; Drug: Oral L-arginine aspartate administration
- the Orn Group (Experimental): Patients received oral L-ornithine aspartate (Farmak, Ukraine) at a dose of 3 g t.i.d. for 15 days after conventional periodontal therapy, n=25.
  Interventions: Procedure: Scaling and root planing; Drug: Oral L-ornithine aspartate administration

INTERVENTIONS:
Procedure: Scaling and root planing — Conventional periodontal therapy, non-surgical periodontal therapy
  Other Names: SRP
Drug: Oral L-arginine aspartate administration — The use of L-arginine aspartate as adjuncts to local conservative treatment (scaling and root planing) of periodontitis to optimize treatment by modulating local macrophage subpopulations
  Other Names: Oral supplementation with Tivortin® Aspartate (Yuria-Pharm, Ukraine)
  Arms: the Arg Group
Drug: Oral L-ornithine aspartate administration — The use of L-ornithine aspartate as adjuncts to local conservative treatment (scaling and root planing) of periodontitis to optimize treatment by modulating local macrophage subpopulations
  Other Names: Oral supplementation with Larnamin (Farmak, Ukraine)
  Arms: the Orn Group

SUMMARY:
The aim of the study was to investigate whether oral administration of L-arginine or L-ornithine could modulate local representation density and ratio of macrophages in periodontitis-affected gingiva by using immunohistochemical detection of CD68+ and CD163+ macrophages in biopsies of the gingiva.

The null hypothesis tested was that L-arginine and L-ornithine have no influences on CD68+ and CD163+ macrophages densities when supplementing the treatment of periodontitis.

Materials and methods. 75 individuals with a diagnosis of generalized periodontitis at stages II-III and grade B (38 women and 37 men, 51% and 49%, respectively) were included in the study. Periodontitis was diagnosed by using the criteria of the Classification of Periodontal and Peri-Implant Diseases and Conditions 2017. 25 patients received scaling and root planing only; 25 patients additionally received L-arginine, and 25 - L-ornithine, according to instructions available in Ukraine.

For the immunohistochemical study of paraffin-embedded sections, the gingival biopsy was taken from 5 selected patients per group before treatment and after 1 month. CD68+ (cluster of differentiation 68 positive) and CD163+ cells served as a morphological equivalent of M1, M2 macrophages subpopulations, and their densities were calculated per 10000 μm2. Statistical analysis was performed by adequate power methods.

DETAILED DESCRIPTION:
Study design The present work was the original research study. 75 individuals with a diagnosis of generalized periodontitis at stages II-III and grade B (38 women and 37 men, 51% and 49%, respectively) were included in the study. Periodontitis was diagnosed by using the criteria of the Classification of Periodontal and Peri-Implant Diseases and Conditions 2017. Stage II of periodontitis was diagnosed in the presence of 3 to 4 mm interdental CAL at the site of greatest loss, 4 to maximum 5 mm PPD, the radiographic bone loss at the root coronal third, and no tooth loss due to periodontitis. Stage III was diagnosed in the presence of ≥5 mm interdental CAL, the radiographic bone loss extending to the middle or apical third of the root, ≤4 teeth loss due to periodontitis. In all cases, periodontitis had a generalized pattern (>30% of teeth involved) and grade B as patterns of the progression, based on indirect evidence (radiographic bone loss expressed as a percentage of root length divided by the age of the subject was from 0.25 to 1.0).

Patients were grouped by stratified randomization into three groups: the SRP Group (patients received scaling and root planing as a full-mouth procedure, n=25); the Arg Group (patients received oral L-arginine aspartate (Yuria-Pharm, Ukraine) at a dose of 1 g t.i.d. for 10 days after SRP, n=25); and the Orn Group (patients received oral L-ornithine aspartate (Farmak, Ukraine) at a dose of 3 g t.i.d. for 15 days after SRP, n=25). We used arginine and ornithine according to instructions for these medicines available for use in Ukraine. During the study, all patients were on a stable diet, without changing their rations and regiments.

For all participants, gender and age were recorded, and periodontal parameters such as periodontal pocket depth (PPD), clinical attachment level (CAL) and bleeding on probing (BoP) measurements were taken from six periodontal sites on all teeth (except for the third molars) by a single calibrated examiner using a manual periodontal probe (dental explorer tool labeled 0106.DT06.CP10, Den Tag, Italy). PPD and CAL were measured to the nearest 1 mm.

All patients were clinically examined before treatment and after 1 month ± 5 days.

Collection of gingival tissue samples For the precise immunohistochemical study, the gingival biopsy of approximately 3x3 mm was excised under local anesthesia before treatment and 1 month later in 5 selected patients per group. Biopsies were obtained in the same time-points, from a single site displaying the deepest pocket around suitable dental and periodontal procedures. Removal of these tissue biopsies did not interfere with the initial treatment plan or influence upon the expected clinical outcomes. After collection, biopsies were fixed in a 4% formalin solution for 24 hr of fixation, dehydrated, and embedded in paraffin.

Immunohistochemistry and antibodies Paraffin sections, 2-3 μm in thickness were deparaffinized and dehydrated. Heat-induced epitope retrieval in citrate buffer, power of hydrogen (pH) 6, was performed by successive heating the slides in the microwave oven, then allowed to cool, rinsed with phosphate-buffered saline (PBS), incubated with blocked reagent, rinsed, and incubated with mouse monoclonal CD68 antibodies (1:30, clone PG-M1, Diagnostic BioSystems, The Hague, The Netherlands) or anti-CD163 (1:100, clone 10D6, Diagnostic BioSystems, The Hague, The Netherlands). Then sections were stained with the 2-steps Mouse/Rabbit PolyVue Plus™ HRP/DAB Detection System (Diagnostic BioSystems, The Hague, The Netherlands), and counterstained with Mayer's haemalaun. PBS was used as a negative control, the lymph node tissue - as a positive control.

Evaluation of immunohistochemical staining CD68+ and CD163+ macrophages (Mφs) were estimated by counting the number of the cells by light microscope ×400 in intensive infiltrative areas, 5 regions from each slice were selected, and all 5 counts were taken for statistics. We counted immunopositive Mφs in the areas of cell infiltration, since they are directly related to inflammation. The number of cells per 10 000 μm2 was calculated as immunopositive cell density. Photos were obtained using the light microscope Axio Lab.A1 (Carl Zeiss, Göttingen, Germany) (×400).

Statistical analysis Small sample size was justified by the expectation of a high effect size, unknown null distribution, and compensated with adequate power non parametric statistics. Precise sample size calculation was not performed.

Means of PPD and CAL were calculated for sites with PD>4mm (affected sites). Statistical analysis was performed using GraphPad Prism 5 software (GraphPad Software, San Diego, USA) by means of descriptive statistics, chi-square test, one-way ANOVA and nonparametric ANOVA tests for multiple comparisons: Friedman - for dependent variables, Kruskal-Wallis test - for independent variables, with post-hoc analyzing. For descriptive statistics of cells numbers, the percentile ranges were also used because of non-normal distributions. The CD68+/CD163+ ratio was assessed by inter-group t-tests comparisons and Spearman correlation checking. P values of <0.05 were considered statistically significant in all of the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Presence of periodontitis
* Good general health
* At least 19 remaining teeth
* Written informed consent forms

Exclusion Criteria:

* Antibiotics or anti-inflammatory medications use within the preceding 3 months
* Periodontal therapy within the previous 6 months
* Purulent exudation from periodontal pockets
* Pregnancy and breastfeeding
* Presence of severe, uncontrolled (decompensated) diseases of the internal organs, or neuropsychiatric disorders
* Presence of other conditions that determined the inability of the patient to understand the nature and possible consequences of the study

Ages: 25 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Periodontal pocket depth (PPD) | Before treatment and after 1 month ± 5 days.
  Mean changes in probing depth (PD). Measurements were taken from six periodontal sites on all teeth (except for the third molars) by a single calibrated examiner using a manual periodontal probe (0106.DT06.CP10, Den Tag, Italy) to the nearest 1 mm.
Clinical attachment level (CAL) | Before treatment and after 1 month ± 5 days.
  Mean changes in clinical attachment level.Measurements were taken from six periodontal sites on all teeth (except for the third molars) by a single calibrated examiner using a manual periodontal probe (0106.DT06.CP10, Den Tag, Italy) to the nearest 1 mm.
Bleeding on probing (BoP) measurements | Before treatment and after 1 month ± 5 days.
  Mean changes in BoP

SECONDARY OUTCOMES:
CD68+ and CD163+ macrophages density in gingiva | Before treatment and after 1 month ± 5 days.
  The number of cells per 10 000 μm2 was calculated as immunopositive cell density

CONTACTS AND LOCATIONS:
Overall Officials: Igor P Kaydashev, Dr.hab., Principal Investigator — Ukrainian Medical Stomatological Academy
Locations (1):
- Ukrainian Medical Stomatological Academy, Poltava, Ukraine

IPD SHARING:
Plan to Share IPD: No
Because all the necessary participant data will be provided in the publication about the study

REFERENCES:
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490
- [Background] Shinkevich VI, Kaidashev IP. [The role of immune cells factors in the remodeling of gingiva at chronic generalized periodontal disease]. Stomatologiia (Mosk). 2012;91(1):23-7. Russian. PMID 22678603
- [Background] Zhou LN, Bi CS, Gao LN, An Y, Chen F, Chen FM. Macrophage polarization in human gingival tissue in response to periodontal disease. Oral Dis. 2019 Jan;25(1):265-273. doi: 10.1111/odi.12983. Epub 2018 Oct 12. PMID 30285304
- [Background] Shynkevych VI, Kaidashev IP. Contribution of macrophage subpopulations to the pathogenesis of chronic periodontitis in humans and perspectives for study. Review of the literature. Zaporozhye medical journal. 2019;21(1): 137-143. doi:10.14739/2310-1210.2019.1.155863.
- [Background] Garaicoa-Pazmino C, Fretwurst T, Squarize CH, Berglundh T, Giannobile WV, Larsson L, Castilho RM. Characterization of macrophage polarization in periodontal disease. J Clin Periodontol. 2019 Aug;46(8):830-839. doi: 10.1111/jcpe.13156. Epub 2019 Jun 25. PMID 31152604
- [Background] Allam JP, Duan Y, Heinemann F, Winter J, Gotz W, Deschner J, Wenghoefer M, Bieber T, Jepsen S, Novak N. IL-23-producing CD68(+) macrophage-like cells predominate within an IL-17-polarized infiltrate in chronic periodontitis lesions. J Clin Periodontol. 2011 Oct;38(10):879-86. doi: 10.1111/j.1600-051X.2011.01752.x. Epub 2011 Aug 31. PMID 21883359
- [Background] Slots J. Periodontitis: facts, fallacies and the future. Periodontol 2000. 2017 Oct;75(1):7-23. doi: 10.1111/prd.12221. PMID 28758294
- [Background] Almubarak A, Tanagala KKK, Papapanou PN, Lalla E, Momen-Heravi F. Disruption of Monocyte and Macrophage Homeostasis in Periodontitis. Front Immunol. 2020 Feb 26;11:330. doi: 10.3389/fimmu.2020.00330. eCollection 2020. PMID 32210958
- [Background] Gordon S, Pluddemann A, Martinez Estrada F. Macrophage heterogeneity in tissues: phenotypic diversity and functions. Immunol Rev. 2014 Nov;262(1):36-55. doi: 10.1111/imr.12223. PMID 25319326
- [Background] Satoh T. [Functional diversity of disorder-specific macrophages]. Rinsho Ketsueki. 2018;59(6):805-811. doi: 10.11406/rinketsu.59.805. Japanese. PMID 29973463
- [Background] Kedia-Mehta N, Finlay DK. Competition for nutrients and its role in controlling immune responses. Nat Commun. 2019 May 9;10(1):2123. doi: 10.1038/s41467-019-10015-4. PMID 31073180
- [Background] Angajala A, Lim S, Phillips JB, Kim JH, Yates C, You Z, Tan M. Diverse Roles of Mitochondria in Immune Responses: Novel Insights Into Immuno-Metabolism. Front Immunol. 2018 Jul 12;9:1605. doi: 10.3389/fimmu.2018.01605. eCollection 2018. PMID 30050539
- [Background] Rath M, Muller I, Kropf P, Closs EI, Munder M. Metabolism via Arginase or Nitric Oxide Synthase: Two Competing Arginine Pathways in Macrophages. Front Immunol. 2014 Oct 27;5:532. doi: 10.3389/fimmu.2014.00532. eCollection 2014. PMID 25386178
- [Background] Nouwen LV, Everts B. Pathogens MenTORing Macrophages and Dendritic Cells: Manipulation of mTOR and Cellular Metabolism to Promote Immune Escape. Cells. 2020 Jan 9;9(1):161. doi: 10.3390/cells9010161. PMID 31936570
- [Background] Hardbower DM, Asim M, Luis PB, Singh K, Barry DP, Yang C, Steeves MA, Cleveland JL, Schneider C, Piazuelo MB, Gobert AP, Wilson KT. Ornithine decarboxylase regulates M1 macrophage activation and mucosal inflammation via histone modifications. Proc Natl Acad Sci U S A. 2017 Jan 31;114(5):E751-E760. doi: 10.1073/pnas.1614958114. Epub 2017 Jan 17. PMID 28096401
- [Background] Moinard C, Caldefie F, Walrand S, Felgines C, Vasson MP, Cynober L. Involvement of glutamine, arginine, and polyamines in the action of ornithine alpha-ketoglutarate on macrophage functions in stressed rats. J Leukoc Biol. 2000 Jun;67(6):834-40. doi: 10.1002/jlb.67.6.834. PMID 10857856
- [Background] Liao SY, Showalter MR, Linderholm AL, Franzi L, Kivler C, Li Y, Sa MR, Kons ZA, Fiehn O, Qi L, Zeki AA, Kenyon NJ. l-Arginine supplementation in severe asthma. JCI Insight. 2020 Jul 9;5(13):e137777. doi: 10.1172/jci.insight.137777. PMID 32497023
- [Background] Simsek B, Cakatay U. Could ornithine supplementation be beneficial to prevent the formation of pro-atherogenic carbamylated low-density lipoprotein (c-LDL) particles? Med Hypotheses. 2019 May;126:20-22. doi: 10.1016/j.mehy.2019.03.004. Epub 2019 Mar 9. PMID 31010493
- [Background] Campion D, Giovo I, Ponzo P, Saracco GM, Balzola F, Alessandria C. Dietary approach and gut microbiota modulation for chronic hepatic encephalopathy in cirrhosis. World J Hepatol. 2019 Jun 27;11(6):489-512. doi: 10.4254/wjh.v11.i6.489. PMID 31293718
- [Background] Ito N, Seki S, Ueda F. Effects of Composite Supplement Containing Collagen Peptide and Ornithine on Skin Conditions and Plasma IGF-1 Levels-A Randomized, Double-Blind, Placebo-Controlled Trial. Mar Drugs. 2018 Dec 3;16(12):482. doi: 10.3390/md16120482. PMID 30513923
- [Background] Fabriek BO, Dijkstra CD, van den Berg TK. The macrophage scavenger receptor CD163. Immunobiology. 2005;210(2-4):153-60. doi: 10.1016/j.imbio.2005.05.010. PMID 16164022